CLINICAL TRIAL: NCT02330640
Title: A Single-center, Prospective,Randomized Study of Antiplatelet Effects of Ticagrelor Versus Clopidogrel in Patients With Dual Anti-platelet Therapy After Coronary Artery Bypass Grafting
Acronym: ATCCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Zhe zheng, Cardiovascular Surgeon Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zzheng
Record Dates: First submitted 2014-12-24; First posted 2015-01-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Antiplatelet Therapy of Coronary Artery Bypass
Keywords: CABG; antiplatelet therapy; ticagrelor
MeSH Terms: interventions — Ticagrelor; Clopidogrel; acetylsalicylic acid lysinate

STUDY DESIGN:
Intervention Model Description: Single center prospective randomized controlled study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ticagrelor (Experimental): 90mg Bid for 30days after first dose
  Interventions: Drug: ticagrelor
- clopidogrel (Active Comparator): 75mg Qd for 30days first dose
  Interventions: Drug: clopidogrel
- asprin (Other): 100mg Qd all patients will be given asprin 100mg Qd within 24hours after CABG
  Interventions: Drug: asprin

INTERVENTIONS:
Drug: ticagrelor — After the operation, the subjects will be randomized into two groups according to the proportion of 1:1; and receive the treatment of aspirin 100mg qd+ticagrelor 90mg bid or the treatment of aspirin 100mg qd+ clopidogrel 75mg qd. The study will plan to enroll 140 subjects in 12 months and the treatment will last for 30 days.
  Arms: ticagrelor
Drug: clopidogrel — After the operation, the subjects will be randomized into two groups according to the proportion of 1:1; and receive the treatment of aspirin 100mg qd+ticagrelor 90mg bid or the treatment of aspirin 100mg qd+ clopidogrel 75mg qd. The study will plan to enroll 140 subjects in 12 months and the treatment will last for 30 days.
  Arms: clopidogrel
Drug: asprin — All patients will be given asprin 100mg Qd within 24hours after operation,and will continue taking aspirin at the end of the study
  Arms: asprin

SUMMARY:
This study is designed to demonstrate that the onset of the antiplatelet effect of 90mg bid dose ticagrelor is more rapid and greater than 75 mg qd dose clopidogrel in patients undergoing CABG surgery.

DETAILED DESCRIPTION:
Patients undergoing coronary artery surgery routinely receive aspirin therapy, as a standard treatment for preserving bypass graft patency. Although the dual antiplatelet therapy post CABG has not been recommended by guideline, present studies indicated the patients could benefit from the dual anti-platelet therapy. Using clopidogrel+aspirin could significantly reduce the early saphenous vein graft occlusion. . Many surgeons empirically prescribe dual anti-platelet therapy in spite of the indeterminacy of the clinical effects. ticagrelor is a novel, reversibly binding, oral, direct-acting P2Y12-receptor antagonist. The ONSET/OFFSET Study also shows that ticagrelor achieved much rapid and greater platelet inhibition than high-loading-dose clopidogrel in patients with stable CAD. ticagrelor is a novel, reversibly binding, oral, direct-acting P2Y12-receptor antagonist. The ONSET/OFFSET Study also shows that ticagrelor achieved much rapid and greater platelet inhibition than high-loading-dose clopidogrel in patients with stable CAD.

ELIGIBILITY:
Inclusion Criteria:

* Female and/or male and ≥ 18 and <80 years of age
* Isolated CABG for the first time
* either on- or off- pump

Exclusion Criteria:

* Combined valvular surgery.
* A second surgery.
* Emergency surgery (a selective operation which change to emergency surgery in some special medical condition).
* Serum creatinine>130μmol/L.
* Oral clopidogrel therapy stops less than 5 days before the surgery.
* Oral anti-coagulation therapy (warfarin) that cannot be withheld.
* History of gastrointestinal or vaginal bleeding, Active pathological bleeding (e.g. active gastroduodenal ulcer or cerebral haemorrhage), history of postoperative gastrointestinal bleeding.
* Uric acid nephropathy, history of postoperative gastrointestinal bleeding.
* History of cerebral haemorrhage.
* Any other condition that may influence platelet count and function.
* Postoperative chest drainage > 200 ml/hr for two hours and more, re-operation for bleeding with persistent cardiac tamponade.
* Treated with IABP or ECMO after operation.
* Any other condition that may put the patient at risk (e.g., recurrent ventricular arrhythmias, peri-operative myocardial infarction, cancer).
* Contraindication to aspirin, clopidogrel and ticagrelor or other reason that study drug should not be administered (e.g., hypersensitivity, moderate or severe liver disease).
* Previous enrollment in other investigational drug or device study within 30 days.

Being or planning to pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
IPA at 2hours | 2 hours after the first dose of study drug
  the platelet inhibition (IPA %) measured by light-transmittance aggregometry at 2 hour in CABG patients after the first dose of study drug

SECONDARY OUTCOMES:
the inhibition of platelet function (IPA%) measured by LTA at 0h, 8h, 24h, 3day, and 30day after the first dose of study drug | 0h, 8h, 24h, 3day, and 30day after the first dose of study drug
  the platelet inhibition (IPA %) measured by light-transmittance aggregometry at 0h, 8h, 24h, 3day, and 30day after the first dose of study drug
the platelet reactivity index at 0h, 2h, 8h, 24h，3day, and 30days | 0h, 2h, 8h, 24h，3day, and 30day after the first dose of study drug
  the platelet reactivity index measured by corrected mean fluorescence intensities (MFIc) at 0h, 2h, 8h, 24h，3day, and 30day after the first dose of study drug in CABG patients.

OTHER OUTCOMES:
The Number of Bleeding events according to BARC definition. | 30 days after the operation
  All the bleeding events will be recorded with BARC definition type1-type5. Considering the specificity of operation, the BARC type1 or type2 bleeding events will not be recorded in the early period of post-operation (7days).
The number of MACE events including all-cause mortality， myocardial infarction, urgent re-operation for heart, cerebral infarction, cerebral hemorrhage. | 30 days after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- FuWaiHospital, Beijing, Beijing Municipality, China